CLINICAL TRIAL: NCT05006170
Title: Pharmacokinetics, Safety, and Efficacy of Dolutegravir Dispersible Tablets in Young Children Living With HIV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTGkids
Record Dates: First submitted 2021-08-04; First posted 2021-08-16 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-07

CONDITIONS: Pediatric HIV Infection
Keywords: dolutegravir dispersible tablet; pharmacokinetics; weight below 20 kg
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Intervention Model Description: Each participants will undergo ARTs medication switch to DTG dispersible tablet, and ABC/3TC dispersible tablet
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 6 to below 10 kg weight band (Experimental): Children with perinatal HIV infection whose weight from 6 kg to below 10 kg
  Interventions: Drug: DTG DT 20 mg
- 10 to below 14 kg weight band (Experimental): Children with perinatal HIV infection whose weight from 10 kg to below 14 kg
  Interventions: Drug: DTG DT 20 mg
- 14 to below 20 kg weight band (Experimental): Children with perinatal HIV infection whose weight from 14 kg to below 20 kg
  Interventions: Drug: DTG DT 25 mg

INTERVENTIONS:
Drug: DTG DT 20 mg — Give 2 tabs of MYLTEGA DT (10mg) PO once daily
  Other Names: MYLTEGA Dispersible Tablet
  Arms: 10 to below 14 kg weight band; 6 to below 10 kg weight band
Drug: DTG DT 25 mg — Give 2.5 tabs of MYLTEGA DT (10mg) PO once daily
  Other Names: MYLTEGA DT Dispersible Tablet
  Arms: 14 to below 20 kg weight band

SUMMARY:
The purpose of this study is to evaluate steady-state pharmacokinetics of DTG dispersible tablets in children with HIV infection weighing from 6 to below 20 kg and to determine the dose of DTG that achieves adult target PK parameter(trough concentration; AUC24h)

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all legal guardians giving written informed consent will undergo check eligibility to enroll the study entry. Patients will be sort into 3 weight band groups 6 to below 10 kg, 10 to below 14 kg, and 14 to below 20 kg. ARTs will be switched to DTG dispersible tablet and ABC/3TC once daily will be prescribed according to weight band dosage. Total of 7 time point of blood sampling for plasma DTG concentrations will be measure at 7-14 day after medication switch. Patient will be follow up as schedule for total 24 week to assess safety, and efficacy of DTG dispersible tablet combine with ABC/3TC.

ELIGIBILITY:
Inclusion Criteria:

* Children living with HIV weighing 6 to below 20 kg
* Naïve to integrase inhibitors

Exclusion criteria:

* Currently active opportunistic infection
* Liver dysfunction (SGPT below 100 IU/mL)
* Renal dysfunction (GFR below 60 mL/min)
* Currently using medication that interacts with DTG

Ages: 3 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Steady-state pharmacokinetics of DTG dispersible tablets in children with HIV infection | At 7-14 day after started on DTG
  Trough plasma DTG concentration and DTG exposure (AUC24h)

SECONDARY OUTCOMES:
Serious adverse event incidence | 24 week after medication switched
  Incidence of grade 3 and 4 adverse events in use of DTG for HIV treatment in
Antiretroviral activity of dolutegravir dispersible tablets combined with two standard background therapies | 24 week after medication switched
  HIV VL <40 copies/mL

CONTACTS AND LOCATIONS:
Overall Officials: Athiporn Premgamone, MD, Principal Investigator — Chulalongkorn University; Thanyawee Puthanakit, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Division of Infectious disease, Department of Pediatrics, Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No